CLINICAL TRIAL: NCT07237009
Title: Effects of Personalized Reminiscence Sessions Delivered by a Digital Conversational Agent to Patients With Neurocognitive Disorders
Brief Title: Effects of Personalized Digital Reminiscence Therapy on Patients With Neurocognitive Disorders
Status: Recruiting | Type: Observational
Sponsor: KompanionCare SAS (Industry)
Collaborators: Clinical Research Units Hungary (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A01382-47_PROTOCOLE_v3.0
Record Dates: First submitted 2025-09-24; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Neurocognitive Disorders, Mild; Cognitive Impairment, Mild; Depression Mild; Apathy; Apathy in Dementia
Keywords: Mild Cognitive Impairment; Dementia; Apathy; Mild Depression; Digital Reminiscence therapy; personalized Reminiscence therapy
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction; Lethargy; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DRT Users: Single observational cohort exposed to a personalized digital reminiscence therapy, through daily 10-15 minute sessions.

SUMMARY:
This study aims to observe the effects of daily personalized digital reminiscence sessions, conducted with the help of a digital conversational agent, and to determine whether these sessions lead to improvements in symptoms such as apathy and depression.

The researchers therefore seek to observe whether this daily use can improve certain aspects of well-being, such as motivation, mood, sleep quality, quality of life, and engagement with the tool.

The study also aims to assess whether simple reminders delivered via the application are sufficient to encourage regular use without external assistance.

Participants will:

* Use the reminiscence app for 25 days for 10-15 minutes.
* Have a primary caregiver help personalize the app by sharing family memories, other relatives may optionally contribute in a private group.
* Complete brief questionnaires at the start and during follow-up routine visits (for example, apathy and depression scales, sleep, and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 60 years of age.
* DSM-5 diagnosis: Early stage of major neurocognitive disorders or MCI (Mild Cognitive Impairment) including all underlying causes.
* Have a Mini-Mental State Exam score of 21 ≤ MMSE ≤ 26.
* Presence of mild depression, or presence of mild apathy, or presence of both
* Displays the necessary physical and cognitive abilities, without major limitations compromising interaction with the digital tool.
* Having voluntarily and informedly agreed to participate in the study (signed written consent).
* Subject's ability to hear and see the digital tool's stimuli (tests integrated into the tool).
* Patients with access to an Apple device (smartphone or tablet), either personal or provided by the sponsor, running iOS version 16 or higher, with internet access.
* Patient has at least one close referent who declares their wish to contribute to the collection of biographical information via the digital messaging group.
* Subjects covered by a social security scheme.

Exclusion Criteria:

* Patients with moderate or severe dementia (MMSE score ≤ 20) because implicit memory recall is less effective in moderate or severe stages for people with PWD.
* Presence of major psychiatric disorders (e.g., schizophrenia, moderate to severe major depressive episode, bipolar disorder).
* Major hearing or visual impairments.
* History of premorbid intellectual disability.
* Patients under guardianship, conservatorship, or legal protection.
* Patients who have already used the Lilia app
* Participating simultaneously in another study involving human subjects, a clinical investigation, or a therapeutic trial for the entire duration of the study.
* Patients who have received a new treatment related to neurocognitive disorders (medication or other) during the 3 months prior to the inclusion visit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited during routine visits at five French university hospital geriatrics/memory clinics.
  The source population comprises older adults followed in these services who live mainly at home or in hospital-based residential settings. The study focuses exclusively on patients with mild neurocognitive disorder or mild dementia, and includes individuals with mild depression.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Baseline, Day 25, Day 50.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated scale of depressive symptom severity.
  Possible scores range from 0 to 60, with higher scores indicating more severe depression.
  Decrease of MADRS total score between two measurement points indicates improvement over time.
  Unit of Measure: points (from 0 to 60)
Change in Lille Apathy Rating Scale (LARS) Total Score | Baseline, Day 25, Day 50.
  The Lille Apathy Rating Scale (LARS) is a clinician-rated questionnaire assessing apathy with a total score from -36 to +36. Higher scores indicating greater apathy. Decrease of LARS total score between two measurement points indicates improvement over time.
  Unit of Measure: points (from -36 to +36).

SECONDARY OUTCOMES:
Change in The Short Form Survey (SF-36) Global Score. | Baseline, Day 25, Day 50.
  The Short Form Survey (SF-36) measures health-related quality of life. Scores range from 0 to 100, with higher scores indicating better health status. Increase of SF-36 global score between two measurement points indicates improvement over time.
  Unit of Measure: Points on SF-36 scale from 0 to 100.
Change in Pittsburgh Sleep Quality Index (PSQI) Global Score | Baseline, Day 25, Day 50.
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire evaluating sleep quality with scores from 0 to 21, with higher scores indicating worse sleep quality. Decrease of PSQI global score between two measurement points indicates improvement over time.
  Unit of Measure: Points on PSQI scale from 0 to 21.
Number of Sessions Completed | From Baseline to Day 25
  Counting the number of sessions completed by the patient between Baseline and Day 25. Higher numbers are indicating greater adherence to the application use.
  Unit of Measure: Number of Sessions Completed
Average Self-Reported Session Duration | From Baseline to Day 25.
  Average self-reported session duration is the approximate average time spent per session with using the Lilia application between Baseline and Day 25 based on the patients' own observations. It is measured by a dedicated question: "On average, how much time did you spend with Lilia when you used it?" (response options: "Less than 5 minutes," "5-10 minutes," "More than 10 minutes").
  Higher values refers to longer average sessions. Unit of Measure: average minutes per session

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Annweiler, Geriatrician, PhD neuroscience, Study Chair — Angers University Hospital Center
Locations (5):
- France (5):
  - CHU Angers, Service médecine gériatrique., Angers
  - Limoges University Hospital Center - Dupuytren Hospital], Geriatric medicine department, Limoges
  - Centre Hospitalier Universitaire de Nice - Institut Claude Pompidou, Centre Mémoire de Ressources et de Recherches (CM2R), Nice
  - APHP Hôpitaux universitaires Paris centre., Paris
  - CHU DE TOURS, Pôle Vieillissement, Hôpital Bretonneau., Tours

IPD SHARING:
Plan to Share IPD: Undecided